CLINICAL TRIAL: NCT05480345
Title: Significance of Impedance Cardiography and Early Repolarization Pattern in Electrocardiogram in Congestive Heart Failure
Brief Title: Significance of Impedance Cardiography and Early Repolarization Pattern in ECG in Congestive Heart Failure
Acronym: SICERE-CHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Andrius Ališauskas, Doctor of Medicine, Assistant lecturer, Lithuanian University of Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HF-ER-001
Record Dates: First submitted 2022-04-06; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Congestive Heart Failure; Chronic Heart Failure; Right Ventricular Failure; Heart Failure
Keywords: Cardiography, impedance; Early repolarization pattern; Electrocardiography; Prognosis
MeSH Terms: conditions — Heart Failure | interventions — Cardiography, Impedance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Impedance cardiography (Experimental): Impedance cardiography parameters recorded with ICG monitor (niccomoTM; Medis, Ilmenau, Germany)
  Interventions: Diagnostic Test: Impedance cardiography

INTERVENTIONS:
Diagnostic Test: Impedance cardiography — Transthoracic impedance cardiography recorded with ICG monitor (niccomoTM; Medis, Ilmenau, Germany): electrodes attached to both sides of the patient's neck (4 electrodes in total) and along the midaxillary line of the left and right sides of the chest (4 electrodes in total), employing the xyphoid process as a reference line.
  Other Names: ICG monitor (niccomoTM; Medis, Ilmenau, Germany)

SUMMARY:
Congestive heart failure (CHF) is a disorder of the heart when structural or functional heart disease impairs the heart's ability to work properly. In developed countries, the prevalence of CHF in the general population is around 1-2% (depending on the definition used) and the prevalence of CHF in people aged 70 years and older is ≥ 10%. The cumulative 5-year mortality of patients with CHF is about 50%.

According to different studies, the prevalence of the early repolarization pattern (ERP) in the 12-lead electrocardiogram (ECG) in the general population is 2-31%. Although ERP in ECG have been considered as benign finding for many years, an increasing number of studies have been conducted in recent years to demonstrate an association of ERP in ECG with sudden cardiac death, mainly through ventricular arrhythmias in previously healthy individuals or those with structural cardiac pathology. New studies are also being performed to support the association of ERP with the progression of CHF.

Although the prevalence of ERP in the general population is not very high, the knowledge that ERP lead to a higher risk of sudden cardiac death and development of CHF lets physicians tailor patient care and follow-up, and treatment at a very low cost because ECG is a cheap, simple, and widely available diagnostic test.

Impedance cardiography (ICG) is another safe, non-invasive, cheap, routine diagnostic method based on the detection of changes in thoracic bioimpedance during heartbeat.

The aim of the present study is to evaluate the diagnostic and prognostic significance of ICG and ERP in congestive heart failure patients and to compare it with other non-invasive CHF diagnostic methods. The investigators hypothesize that ERP and changes in ICG readings may be used as a cheap, safe, non-invasive and widely available diagnostic and prognostic methods in patients with congestive heart failure witch help physicians tailor their patient follow-up and treatment accordingly.

The participants of the study are those who are hospitalized due to the flare-up of congestive heart failure. All of the participants will undergo routine tests. They will also undergo an ICG witch is not a routine test in the research center.

DETAILED DESCRIPTION:
Congestive heart failure (CHF) is a disorder of the heart when structural or functional heart disease impairs the heart's ability to fill with blood or pump it out properly. In developed countries, the prevalence of CHF in the general population is around 1-2% (depending on the definition used) and the prevalence of CHF in people aged 70 years and older is ≥ 10%. The cumulative 5-year mortality of patients with CHF is about 50%. In 2018 in Lithuania CHF accounted for 5.64 hospitalizations per 1000 people in general population. Mortality rate was 155.17 per 1,000 patients and the average length of in hospital stay was 26.64 days.

In order to improve the diagnosis, treatment and financial costs in patients with CHF it is important to search for diagnostic methods that are cheap, effective, preferably non-invasive, as well as those that have reliable prognostic significance for patients with CHF.

According to different studies, the prevalence of early repolarization pattern (ERP) in the 12-lead electrocardiogram (ECG) in the general population is 2-31%. This may be due to different ERP definitions used by different authors. Although ERP in ECG have been considered as benign finding for many years, an increasing number of studies have been conducted in recent years to demonstrate an association of ERP in ECG with sudden cardiac death, mainly through ventricular arrhythmias in previously healthy individuals or those with structural cardiac pathology. New studies are also being performed to support the association of ERP in ECG with the progression of CHF. ERP, which has been first described in 1936 by Shipley and Hallaran, is generally defined as J-point (J-p) elevation with QRS notching or slurring in the terminal part of the QRS complex in at least two adjacent inferior (II, III, and aVF) and / or lateral leads (I, aVL, and V4-V6) detected by the standard 12-lead electrocardiogram. The amplitude of the J point must be at least 1 mm (0.1 mV) and the J-p must appear as an additional positive wave in the S wave (QRS notching) or the J-p may appear as a faint transition of the high R wave to the ST segment without Jp-QRS slurring, QRS duration should be <120 ms and anterior precordial leads (V1-3) are not included in the description of ERP because such changes in these leads may be due to Brugada syndrome or right ventricular dysplasia. Although the prevalence of ERP in ECG in the general population is not very high, the knowledge that ERP in ECG lead to a higher risk of sudden cardiac death and development of CHF lets physicians tailor patient care and follow-up, and treatment at a very low cost because an ECG is a cheap, simple, and widely available diagnostic test.

Impedance cardiography (ICG) is another safe, non-invasive, cheap, routine diagnostic method based on the detection of changes in thoracic bioimpedance during heart cycle. A lot of research has been carried out in recent years which examines the possibilities of ICG in CHF patients in various aspects: diagnostics, treatment, prognosis. A good correlation between ICG, cardiac ultrasound and invasive diagnostic methods was observed in most studies.

Evaluating CHF patients, it is important to evaluate thoracic fluid content (TFC) that can be used to diagnose a flare-up of CHF, its degree, to evaluate the effectiveness of treatment, as well as the prognosis of patients. ICG evaluate the TFC and its index. In clinical practice, it is important to predict the flare-ups of CHF, to predict the outcome of CHF patients, and to provide appropriate treatment to patients timely. Various prognostic indicators are studied: ICG parameters (TFC, TFC index, cardiac output (CO), CO index, systolic time ratio, etc.), brain natriuretic peptide (BNP), New York Heart Association (NYHA) classes. The current data are quite controversial, with most studies reporting positive ICG data as a predictor of CHF.

The aim of the present study is to evaluate the diagnostic and prognostic significance of ICG and ERP in ECG in CHF patients and to compare it with other non-invasive CHF diagnostic methods. The investigators hypothesize that ERP in ECG and changes in ICG readings may be used as a cheap, safe, non-invasive and widely available diagnostic and prognostic methods in patients with CHF witch help physicians tailor their patient follow-up and treatment accordingly.

The participants of the study are those who are hospitalized due to the flare-up of CHF. All of the participants will undergo routine tests. They will also undergo an ICG witch is not a routine test in the research center.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized due to a flare-up of congestive heart failure;
* early repolarization pattern in a 12-lead ECG;
* free from mental disorders;
* participants signed the informed consent form.

Exclusion Criteria:

* septic shock;
* high grade aortic valve regurgitation;
* high grade aortic valve stenosis;
* ventricular septal defect;
* prosthetic aortic valve;
* uncontrolled hypertension (mean arterial pressure >130 mmHg);
* heart rate > 200 bpm;
* height <120 cm or >230 cm;
* weight <30 kg or >155 kg;
* intra-aortic balloon counterpulsation;
* pacemaker with a minute ventilation sensor;
* restless patient;
* patient refuses to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
In-hospital stay duration | Day of discharge from the hospital or day of death from any cause, whichever came first, assessed throughout the whole hospital admission stay
  In-hospital stay duration measured in days: early patient outcomes (discharge time from the hospital or time of any cause death)
Rehospitalizations | Follow-up up to 12 months
  Latter patient outcomes: number of rehospitalizations due to congestive heart failure
Time of death | From date of hospitalization until the date of death of congestive heart failure, follow-up through study completion, an average of 1.5 year
  Latter patient outcomes: time to death (measured in days) due to congestive heart failure. Data were collected from Lithuanian medical record database (Electronic information system's of health services and cooperation infrastructure)

SECONDARY OUTCOMES:
Early patient outcome 1a | On the day of patient's discharge from the hospital
  Early patient outcomes: repeated evaluation of TFC on the day of discharge from the hospital
Early patient outcome 1b | On the day of patient's discharge from the hospital
  Early patient outcomes: repeated evaluation TFC index on the day of discharge from the hospital
Early patient outcome 2a | On the day of patient's discharge from the hospital
  Early patient outcomes: repeated evaluation of cardiac output (CO) on the day of discharge from the hospital
Early patient outcome 2b | On the day of patient's discharge from the hospital
  Early patient outcomes: repeated evaluation of CO index on the day of discharge from the hospital
Early patient outcome 3 | On the day of patient's discharge from the hospital
  Early patient outcomes: repeated evaluation of systolic time ratio (STR) on the day of discharge from the hospital
Early patient outcome 4a | On the day of patient's discharge from the hospital
  Early patient outcomes: repeated evaluation of left cardiac work (LCW) on the day of discharge from the hospital
Early patient outcome 4b | On the day of patient's discharge from the hospital
  Early patient outcomes: repeated evaluation of left cardiac work index (LCWI) on the day of discharge from the hospital
Serum BNP level | On the day of patient's discharge from the hospital
  Serum BNP level on the day of discharge from the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Andrius Ališauskas, MD, Principal Investigator — Lithuanian University of Health Sciences
Locations (1):
- Lithuanian University of Health Sciences Kaunas Hospital, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available from 2022-08-01 through 2027-08-01.
Access Criteria: Data will be shared with other principal investigators in the field of congestive heart failure research. Requests should be submitted to study's principal investigator MD Andrius Ališauskas at: andrius.alisauskas@lsmu.lt